CLINICAL TRIAL: NCT07000643
Title: Proton Therapy Versus Photon Therapy for the Treatment of Nasopharyngeal Carcinoma: A Prospective, Open-Label, Multicenter, Phase III Non-Inferiority Clinical Trial
Brief Title: Phase III Non-Inferiority Trial of Proton Versus Photon Therapy for Nasopharyngeal Carcinoma
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Man Hu (Other)
Responsible Party: Sponsor-Investigator, Man Hu, Chief physician, Shandong Cancer Hospital and Institute
Organization: Shandong Cancer Hospital and Institute (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SDZLEC2025-067-01
Record Dates: First submitted 2025-05-24; First posted 2025-06-03 (Actual); Last update posted 2025-06-03 (Actual); Status verified 2025-02

CONDITIONS: Nasopharyngeal Carcinoma
Keywords: Nasopharyngeal carcinoma; proton radiotherapy; target area delineation
MeSH Terms: conditions — Nasopharyngeal Carcinoma | interventions — Radiotherapy, Intensity-Modulated

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- IMPT Group (Experimental): Patients in this group will receive Intensity-Modulated Proton Therapy (IMPT). The systemic therapy plan will be formulated according to clinical guidelines. These patients have histologically confirmed, previously untreated, non-metastatic (M0) nasopharyngeal carcinoma.
  Interventions: Radiation: Intensity-Modulated Proton Therapy (IMPT)
- IMRT Group (Other): Patients in this group will receive Intensity-Modulated Radiotherapy (IMRT). IMRT is currently one of the most widely used techniques and serves as a standard treatment. The systemic therapy plan will be formulated according to clinical guidelines. These patients have histologically confirmed, previously untreated, non-metastatic (M0) nasopharyngeal carcinoma.
  Interventions: Radiation: Intensity-Modulated Radiotherapy (IMRT)

INTERVENTIONS:
Radiation: Intensity-Modulated Proton Therapy (IMPT) — This is the experimental arm intervention. Patients receive Intensity-Modulated Proton Therapy (IMPT) for primary nasopharyngeal carcinoma.
  The subjects are patients with histologically confirmed, previously untreated, non-metastatic (M0) nasopharyngeal carcinoma.
  Radiotherapy target volumes and doses: GTV (gross tumor volume of primary tumor and metastatic lymph nodes); CTV70Gy (GTVp + 0-5mm margin, GTVn + 0-3mm margin, reducible near organs at risk) at a dose of 69.6-70Gy; CTV50-54Gy (GTVp + 8-10mm margin + entire nasopharyngeal mucosa + adjacent high/intermediate risk structures and intermediate-risk subclinical lymph node regions) at a dose of 50-54Gy, delivered at 2Gy/(RBE) per fraction. The protocol notes that proton therapy does not use a PTV (Planning Target Volume).
  The systemic therapy plan is formulated according to clinical guidelines.
  Arms: IMPT Group
Radiation: Intensity-Modulated Radiotherapy (IMRT) — This is the control arm intervention. Patients receive Intensity-Modulated Radiotherapy (IMRT) for primary nasopharyngeal carcinoma; IMRT is one of the current standard and widely used treatment techniques.
  The subjects are patients with histologically confirmed, previously untreated, non-metastatic (M0) nasopharyngeal carcinoma.
  Radiotherapy target volumes and doses: GTV (gross tumor volume of primary tumor and metastatic lymph nodes); CTV70Gy (GTVp + 0-5mm margin, GTVn + 0-3mm margin); PTV70 (CTV70 + 3-5mm margin, reducible near organs at risk) at a dose of 70Gy; CTV50-54Gy (GTVp + 8-10mm margin + entire nasopharyngeal mucosa + adjacent high/intermediate risk structures and intermediate-risk subclinical lymph node regions); PTV50-54 (CTV50-54 + 3-5mm margin, reducible near organs at risk) at a dose of 50-54Gy, delivered at 2Gy/(RBE) per fraction.
  The systemic therapy plan is formulated according to clinical guidelines.
  Arms: IMRT Group

SUMMARY:
This study is a prospective, open-label, multicenter, cohort, phase III non-inferiority clinical trial comparing proton therapy with photon radiotherapy for nasopharyngeal carcinoma. It intends to enroll histologically confirmed newly diagnosed nasopharyngeal carcinoma patients without distant metastasis (M0). Through a prospective 1:1 matched cohort study design, patients will be divided into the intensity-modulated proton therapy (IMPT) group and the intensity-modulated radiation therapy (IMRT) group. Systemic treatment regimens are formulated according to clinical guidelines.

DETAILED DESCRIPTION:
This is a prospective, open-label, multicenter, cohort, phase III non-inferiority clinical trial comparing proton therapy with photon radiotherapy for nasopharyngeal carcinoma. Histologically confirmed newly diagnosed nasopharyngeal carcinoma patients without distant metastasis (M0) will be enrolled and allocated to the intensity-modulated proton therapy (IMPT) group or intensity-modulated radiation therapy (IMRT) group via a prospective 1:1 matched cohort design. Systemic treatment regimens are formulated according to clinical guidelines.

Study Phase： Phase III Study Endpoints：

Primary Endpoint:

2-year locoregional recurrence-free survival (LRFS).

Secondary Endpoints:

2-year overall survival (OS), 2-year progression-free survival (PFS), 2-year distant metastasis-free survival (DMFS), radiation-related adverse reactions, and quality of life.

Inclusion Criteria：

Patients must meet all the following criteria:

Signed written informed consent before any trial-related procedures; Aged ≥18 and ≤75 years, regardless of gender; Histologically confirmed nasopharyngeal carcinoma, including keratinizing carcinoma, non-keratinizing differentiated carcinoma, and undifferentiated carcinoma (latest WHO classification); Clinically diagnosed as nasopharyngeal carcinoma (cT1-4N0-3M0, AJCC 9th edition); No prior systemic antitumor therapy for locally advanced disease; ECOG performance status 0-1;

Sufficient organ function with the following laboratory parameters:

Absolute neutrophil count (ANC) ≥1.5×10⁹/L; Platelets ≥75×10⁹/L; hemoglobin ≥9 g/dL (90 g/L or ≥5.6 mmol/L); Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤2.5×ULN; Serum creatinine ≤1.5×ULN and creatinine clearance ≥60 ml/min (calculated by Cockcroft-Gault formula); Normal coagulation function and myocardial enzymes without clinical significance.

Exclusion Criteria：

Patients with any of the following will be excluded:

Distant metastasis (M1); Head and neck squamous cell carcinoma originating from non-nasopharyngeal sites; Pathological types other than nasopharyngeal keratinizing carcinoma and non-keratinizing carcinoma; Currently participating in an interventional clinical trial; Contraindications to radiotherapy;

Active hepatitis B infection (defined as HBsAg-positive with HBV-DNA copy number above the upper limit of normal), except:

HBV viral load <1000 copies/ml (200 IU/ml) with anti-HBV therapy throughout the study; Anti-HBc(+), HBsAg(-), anti-HBs(-), and HBV viral load (-) (requires close monitoring for reactivation); Active HCV infection (HCV antibody-positive with HCV-RNA above the lower limit of detection); Pregnant women;

Severe or uncontrolled systemic diseases, such as:

Significant cardiac arrhythmias (e.g., complete left bundle branch block, ≥Grade II heart block, ventricular arrhythmia, atrial fibrillation); Unstable angina, congestive heart failure (NYHA ≥ Class 2); Arterial thrombosis, embolism, or ischemia within 6 months before enrollment; Interstitial lung disease requiring glucocorticoid therapy within 1 year or current active disease; Active tuberculosis; Active or uncontrolled infection requiring systemic treatment; Clinically active diverticulitis, intra-abdominal abscess, gastrointestinal obstruction; Severe liver diseases (e.g., cirrhosis, decompensated liver disease, acute/chronic active hepatitis); Mental disorders precluding study participation; Medical history, diseases, treatments, or laboratory abnormalities interfering with trial results, or other conditions deemed unsuitable by the investigator.

Evaluation Criteria

Efficacy Evaluation:

Primary and secondary endpoints are assessed by investigators according to RECIST 1.1:

LRFS: Time from randomization to locoregional recurrence (primary/lymph node recurrence or death from any cause); OS: Time from randomization to death from any cause; PFS: Time from enrollment to disease progression, recurrence, or death; DMFS: Time from randomization to distant metastasis or death.

Toxicity Assessment:

Acute and late radiation-related adverse reactions (e.g., mucosal/skin reactions, gastrointestinal reactions, myelosuppression, xerostomia, hearing loss) are graded per NCI CTCAE v5.0.

Quality of Life:

Assessed using EORTC QLQ-C30(V3.0) and QLQ-H&N35(V1.0) at baseline, weekly during treatment, post-treatment, and follow-ups.

Safety Evaluation:

Adverse events (AEs), treatment-emergent AEs (TEAEs), serious AEs (SAEs); Proportion of patients discontinuing treatment due to AEs; Changes in vital signs, physical examinations, and laboratory parameters. Statistical Plan and Sample Size

Sample Size Calculation:

Non-inferiority design assuming 2-year LRFS of 85% for IMRT. With one-sided α=0.025, power=0.8, 1:1 ratio, and non-inferiority margin δ=8%, PASS software estimates 193 patients per group (386 total), accounting for 5% loss to follow-up.

Statistical Methods:

Efficacy analyzed in Intention-to-Treat (ITT) and Per Protocol (PPS) populations; safety in Safety Set (SS). Survival curves estimated by Kaplan-Meier, compared by log-rank test. Multivariate analysis uses Cox proportional hazards model. LRFS is one-sided test (α=0.025); others are two-sided (α=0.05).

ELIGIBILITY:
Inclusion Criteria:

Signed written informed consent prior to the implementation of any trial-related procedures; No gender restriction, age ≥18 years and ≤75 years; Histologically confirmed, according to the latest WHO classification, including keratinizing carcinoma, non-keratinizing differentiated carcinoma, and undifferentiated carcinoma; Investigator-assessed nasopharyngeal carcinoma (cT1-4N0-3M0, AJCC 9th Edition); No prior systemic anti-tumor therapy for locally advanced disease; ECOG performance status 0-1;

Adequate organ function, subjects must meet the following laboratory parameters:

Absolute neutrophil count (ANC) ≥1.5x10⁹/L. Platelets ≥75×10⁹/L. Hemoglobin ≥9 g/dL (90 g/L) or ≥5.6 mmol/L; Aspartate aminotransferase (AST) and Alanine aminotransferase (ALT) ≤2.5×ULN (Upper Limit of Normal) Serum creatinine ≤1.5×ULN AND creatinine clearance (calculated using Cockcroft-Gault formula) ≥60 ml/min; Good coagulation function: simple laboratory abnormalities judged by the investigator to be without clinical significance; Myocardial enzyme spectrum: simple laboratory abnormalities judged by the investigator to be without clinical significance; (Note: The document lists this as criteria 8 under 3.2.1 in the main text, but the synopsis table formatting places it slightly differently though it appears to be the last point of item 7 in structure. For clarity, listing as a separate main point as per the detailed protocol structure.)

Exclusion Criteria:

Presence of distant metastatic lesions (M1). Primary squamous cell carcinoma of the head and neck not originating in the nasopharynx.

Diagnosis of types other than nasopharyngeal keratinizing carcinoma and non-keratinizing carcinoma; (Note: The inclusion criteria state WHO types: keratinizing, non-keratinizing differentiated, and undifferentiated. This exclusion seems to narrow it further or implies a nuance. This is a direct translation of the source.) Currently participating in an interventional clinical research treatment; Contraindications to radiotherapy;

Untreated active hepatitis B (defined as HBsAg positive with HBV-DNA copy number greater than the upper limit of normal at the respective study center's laboratory); Note: Hepatitis B subjects meeting the following criteria may also be enrolled:

HBV viral load <1000 copies/ml (200 IU/ml) before the first dose; subjects should receive anti-HBV therapy throughout the study drug treatment period to avoid viral reactivation.

For subjects who are anti-HBc (+), HBsAg (-), anti-HBs (-), and HBV viral load (-), prophylactic anti-HBV therapy is not required, but close monitoring for viral reactivation is necessary.

Active HCV infection (HCV antibody positive and HCV-RNA level above the lower limit of detection); Pregnant women;

Presence of any severe or uncontrolled systemic diseases, for example:

Significant and symptomatically severe, difficult-to-control abnormalities in rhythm, conduction, or morphology on resting electrocardiogram, such as complete left bundle branch block, second-degree or higher heart block, ventricular arrhythmias, or atrial fibrillation[cite: 2]; Unstable angina, congestive heart failure, chronic heart failure of New York Heart Association (NYHA) class ≥ 2; Any arterial thrombosis, embolism, or ischemia within 6 months prior to enrollment, such as myocardial infarction, unstable angina, cerebrovascular accident, or transient ischemic attack[cite: 2]; History of non-infectious pneumonitis requiring glucocorticoid therapy within 1 year prior to the first dose, or currently active interstitial lung disease; Active pulmonary tuberculosis; Active or uncontrolled infection requiring systemic therapy; Clinically active diverticulitis, intra-abdominal abscess, gastrointestinal obstruction; Liver diseases such as severe cirrhosis, decompensated liver disease, acute or chronic active hepatitis; Patients with mental disorders who cannot cooperate with treatment; History of illness or disease, treatment, or abnormal laboratory values that could interfere with study results, hinder the subject's full participation in the study, or other situations deemed unsuitable for enrollment by the investigator; or if the investigator believes there are other potential risks making the subject unsuitable for this study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 386 (Estimated)
Dates: Start 2025-05-07 (Actual); Primary Completion 2027-02-28 (Estimated); Study Completion 2029-02-28 (Estimated)

PRIMARY OUTCOMES:
2-year Locoregional Recurrence-Free Survival (LRFS) | 2 years
  Defined as the time from group allocation to local-regional recurrence, including recurrence at the primary site and lymph node regions, or death from any cause.

SECONDARY OUTCOMES:
2-year Overall Survival (OS) | 2 years
  Time from group allocation to death from any cause
2-year Progression-Free Survival (PFS) | 2 years
  Defined as the time from enrollment to documented disease progression or recurrence, or death from any cause.
2-year Distant Metastasis-Free Survival (DMFS) | 2 years
  Time from group allocation to the occurrence of distant metastasis or death from any cause
Radiation-related adverse reactions | During the study process and follow-up period (acute adverse reactions assessed mainly during treatment and shortly thereafter; late adverse reactions assessed during long-term follow-up according to the follow-up schedule: every 3 months within 2 years,
  The severity of acute and late radiation-related adverse reactions (e.g., mucosal reactions, skin reactions, gastrointestinal reactions, myelosuppression, xerostomia, hearing loss, temporal lobe injury, etc.) will be graded and assessed according to NCI CTCAE Version 5.0
Quality of Life | Before treatment, weekly during treatment, at the end of treatment, and at each follow-up visit (follow-up visits scheduled every 3 months within 2 years, every 6 months between 2 to 5 years, and every 12 months after 5 years ).
  Assessed using the European Organisation for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaires QLQ-C30 (V3.0) and QLQ-H&N35 (V1.0).

CONTACTS AND LOCATIONS:
Overall Officials: Man Hu, Dr, Study Chair — Shandong Cancer Hospital and Institute, Shandong First Medical University and Shandong Academy of Medical Sciences
Locations (1):
- Shandong Cancer Hospital and Institute, Shandong First Medical University and Shandong Academy of Medical Sciences, Jinan, China

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR